CLINICAL TRIAL: NCT04185753
Title: Chronotropic Incompetence During Cardiopulmonary Exercise Testing in Obese Adolescents: Associations With Caridometabolic Health
Brief Title: Chronotropic Incompetence During Exercise Testing in Obese Adolescents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Dominique Hansen, Principal Investigator, Hasselt University
Other Study IDs: CIDCET study
Record Dates: First submitted 2019-11-27; First posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Obesity, Childhood; Cardiac Disease; Cardiovascular Risk Factor
MeSH Terms: conditions — Pediatric Obesity; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese adolescents with CI: Obese adolescents with chronotropic incompetence
  Interventions: Diagnostic Test: The prevalence of chronotropic incompetence during maximal cardiopulmonary exercise testing
- Control group: Obese adolescents without chronotropic incompetence
  Interventions: Diagnostic Test: The prevalence of chronotropic incompetence during maximal cardiopulmonary exercise testing

INTERVENTIONS:
Diagnostic Test: The prevalence of chronotropic incompetence during maximal cardiopulmonary exercise testing — The prevalence of chronotropic incompetence during maximal cardiopulmonary exercise testing

SUMMARY:
In adolescents with obesity cardiopulmonary exercise testing (CPET) has become an important clinical examination providing valuable information with regard to the integrative exercise responses, including the pulmonary, cardiovascular and muscular systems.

During CPET, mechanical constraints in ventilation, an elevated risk for hypoxia and chronotropic incompetence (CI) (defined as the inability of the heart to increase its rate with increased activity), or compromised cardiac function (e.g. lowered heart rate (HR) recovery, chronotropic index and stroke volume) are often observed in obese adults. Moreover, several studies regarding exercise capacity and cardiopulmonary responses to maximal endurance exercise testing have been performed in obese adolescents. Despite these previous investigations in obese adolescents it remains controversial whether cardiopulmonary disturbances can be observed consistently during CPET. However, a number of studies have reported a suboptimal response to exercise, in particular a reduced peak heart rate (HRpeak) and peak cycling power output (Wpeak). Adult obesity modifies cardiac behavior, including resting HR and CI, which has a marked effect on exercise capacity. Therefore, chronotropic variables are the most important factors that affect exercise performance. It has been shown that both peak and resting HR account for over forty percent of variability of exercise capacity. Interestingly, resting HR and HR response to exercise, including a blunted HR increase, low chronotropic index and HR recovery, are important predictors of all-cause mortality and cardiovascular death, at least in adults. These changes in HR during and recovery from CPET are mediated by the balance between sympathetic and vagal activity of the autonomic nervous system. Adverse cardiovascular outcomes associated with the metabolic syndrome may be mediated by autonomic dysfunction, whereby obesity is characterized by sympathetic predominance and a decrease in vagal activity in the basal state, where reduced sympathetic responsiveness has been observed during exercise. Therefore, these multiple exercise risk markers could provide valuable clinical information regarding cardiometabolic health. Nonetheless HR behavior during CPET has not been described in obese adolescents. The goal of this study is to examine the HR behavior of obese adolescents during CPET to clarify whether this population suffer from CI.

ELIGIBILITY:
Inclusion Criteria:

* obese or lean (based on extended international (IOTF) body mass index cut-offs for thinness, overweight and obesity)
* Parental permission

Exclusion Criteria:

* Chronic cardiovascular, renal, pulmonary or orthopaedic disease
* Medication use that could possibly influence the heart rate

Ages: 11 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Obese adolescents
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-11-29 (Estimated); Primary Completion 2020-01-15 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
Heart rate (HR) during exercise testing | day 1
  Assessed using a 12-lead ECG device
Peak oxygen uptake (VO2) during exercise testing | day 1
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VO2 is collected breath-by-breath and averaged every ten seconds.
Peak workload during exercise testing | day 1
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed and the incremental workload is measured

SECONDARY OUTCOMES:
Body height | day 1
  Body height is measured to the nearest 0.1cm using a wall-mounted Harpenden stadiometer, with participants barefoot
Body weight | day 1
  Body weight (in underwear) is determined using a digital-balanced weighting scale to the nearest 0.1kg
Waist circumference | day 1
  Waist circumference will be measured to the nearest 0.1cm using a flexible metric measuring tape with participants barefoot (in underwear) in standing position. Waist circumference is measured at the midpoint between the lower rib margin and the top of the iliac crest.
Hip circumference | day1
  Hip circumference will be measured to the nearest 0.1cm using a flexible metric measuring tape with participants barefoot (in underwear) in standing position. Hip circumference is measured at the widest circumference of the hip at the level of the greater trochanter.
Physical activity questionnaire for adolescents (PAQ-A) | day 1
  physical activity determined using the validated Dutch physical activity questionnaire for adolescents
Tanner stage | day 1
  Puberty stage (ranging from 1 to 5) will be assessed in all participants by the pediatric endocrinologist using Tanner staging criteria.
Plasma glucose | day 1
  Blood analyses
Total cholesterol | day 1
  Blood analyses
High-density lipoprotein cholesterol | day 1
  Blood analyses
Low-density lipoprotein cholesterol | day 1
  Blood analyses
Triglyceride concentration | day 1
  Blood analyses
C-reactive protein | day 1
  Blood analyses
Serum leptin concentration | day 1
  Blood analyses
Insulin | day 1
  Blood analyses
Homeostatic model assessment for insulin resistance (HOMA-IR) | day 1
  Homeostatic model assessment for insulin resistance calculated from insulin and glucose concentration
Carbon dioxide output (VCO2) during exercise testing | day 1
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VCO2 is collected breath-by-breath and averaged every ten seconds.
Minute ventilation(VE) during exercise testing | day 1
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VE is collected breath-by-breath and averaged every ten seconds.
Tidal volume (Vt) during exercise testing | day 1
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis Vt is collected breath-by-breath and averaged every ten seconds.
Breathing frequency (BF) during exercise testing | day 1
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis BF is collected breath-by-breath and averaged every ten seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Hansen, PhD, Principal Investigator — Hasselt University
Locations (1):
- Virga Jesse hospital - Heart centre Hasselt, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No